CLINICAL TRIAL: NCT03191630
Title: Increasing Activity Post-Kidney Transplant With SystemCHANGE
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017B0084; 1K23NR016274-01A1 (NIH)
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-02

CONDITIONS: Kidney Transplant; Complications; Physical Activity; Cardiorenal; Change; Cardiovascular Diseases
Keywords: Kidney transplant; SystemCHANGE; physical activity; smart phone; Fitbit; activity monitor; step count; post-surgery; quality of life; cardiovascular
MeSH Terms: conditions — Motor Activity; Cardiovascular Diseases | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Participants in the intervention group will receive the combination of the SystemCHANGE and activity tracker intervention while participants in the control group will use activity trackers only. Intervention and control groups will receive the same instruction on use of the activity tracker, and have the same number of study contacts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): This arm includes participants randomized to the control group who will use activity trackers (Fitbits) only, and not receive the SystemCHANGE intervention.
  Interventions: Behavioral: Fitbit (Control)
- Intervention (Experimental): This are includes participants randomize to the intervention group who will receive the combination of the SystemCHANGE TM and activity tracker intervention
  Interventions: Behavioral: SystemCHANGE and Fitbit (Intervention)

INTERVENTIONS:
Behavioral: Fitbit (Control) — Study procedures include group sessions at the OSU Transplant Clinic with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12. Session 1 for the control group will be identical to the Intervention with the only exception being that participants in the control group will not be asked to increase their step goal. Throughout their participation, subjects will be asked questions only about their use of the Fitbit activity tracker. The research team will not be in contact with them for 6 months, after which time there will be a final group session.
  Other Names: Fitbit
  Arms: Control
Behavioral: SystemCHANGE and Fitbit (Intervention) — Study procedures include group sessions with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12. Study personnel will demonstrate proper Fitbit activity tracker use, and teach participants to sync to their smartphone and retrieve data from their Fitbit. Subjects will be called to encourage them to increase their step goal 5% each month. Fitbit activity tracker reports will be reviewed and participants will be asked to identify what people or things influence their physical activity. Subjects will be asked what they are learning about physical activity, their contentment level with current physical activity, and if they want to make changes. Participants will continue for months, after which time there will be a final group session.
  Other Names: SystemCHANGE and Fitbit
  Arms: Intervention

SUMMARY:
Inactivity is a common problem among older kidney transplant recipients (KTRs) and is associated with their high incidence of obesity and cardiovascular problems which are the leading cause of death for KTRs. However, the combination of SystemCHANGE activity trackers holds promise for increasing physical activity of KTR patients post-surgery.

This pilot study will incorporate Fitbit health trackers with an intervention of questions about influences to physical activity in a population of kidney transplant recipients who are at particularly high risk of cardiovascular disease and death.

DETAILED DESCRIPTION:
This is a randomized study with intervention and control arms of sixty kidney transplant recipients age 60 and older. Demographic information will be collected during the screening phone call and will include: gender, race, marital status, income, education, transplant date, prescribed medications, type of diet, smoking status, and co-morbidities. All study data will be entered directly into electronic research forms using REDCap.

Overview of Intervention and Control Groups:

Intervention and control groups will be enrolled in the study in the same manner, receive the same instruction on use of the Fitbit and have the same number of study contacts. Group sessions will be held at the OSU Transplant Clinic with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12.

Intervention Group Active Phase, Group Session 1 (1 hour, 20 minutes): Research staff will demonstrate proper Fitbit activity tracker use, set up the smartphone application, and assist entry of daily step goals into the smartphone application. Fitbits will be set up with Gmail accounts with unique unidentifiable codes. Participants will be taught how to sync to their smartphone and retrieve data from their Fitbit. One week following this session, participants will be called to troubleshoot problems and be encourage to increase their step goal 5% each month (total phone time 15 minutes).

Intervention/Control Group Timeline:

Intervention Active Phase, Group Session 2 (1 hour): Fitbit activity tracker reports will be reviewed by research staff with participants. SystemCHANGE concepts will be discussed such as "opportunities for improvement" and "possibilities for doing better."

A SystemCHANGE powerpoint will outline components and participants will be placed in groups of 5 where researchers will guide participants through the 4 steps of SystemCHANGE.

Participants will be asked to identify important people that influence their physical activity, which habits or activity occur daily, weekly, or monthly, and how these habits and people impact physical activity. Participants will also include things that influence their participation in physical activity (e.g., availability of facilities as a walking path getting home from work late, or sleeping late on a weekend). Social activities and any rituals associated with physical activity such as gardening, housecleaning, shopping, and hobbies will also be noted. Research staff will place the routines (daily, weekly, monthly) into a graphic format that helps participants understand how routines are related to each other and can work for, or against, changing physical activity behavior. These cycles will be discussed to help understanding of how a routine involving family demands, for example, may influence participation in physical activity. Goals for increasing steps will be made, (generally, a 5% increase) and use of their activity tracker reports for monitoring progress toward improvement will be discussed and demonstrated. In this session and throughout, participants will be encouraged to look beyond personal motivation and explore their life routines and the people who shape those routines.

Intervention Active Phase, Group Sessions 3-7 (1 hour/session): Prior to each session, the participants' activity tracker reports will be given to them and reviewed during the group session. Participants will be asked what they are learning about their physical activity and what changes they want to make. Participants will be asked to describe their improvements and be encouraged to continue using the activity tracker for the next 6 months during the maintenance phase.

Intervention Maintenance (6 months): At the final monthly session, participants will be instructed to continue until month 12.

Control Group Session 1 for the control group will be identical to the Intervention with the only exception being that participants in the control group will NOT be asked to increase their step goal 5% each month based on the step-data received from baseline to week 1.

Session 2 will be used to troubleshoot and discuss any problems with the Fitbit activity trackers. In later sessions, educational information about healthy living as a transplant recipient will be presented, including topics such as diet, taking medication, risk for skin cancer, gastrointestinal side effects, dental care, and new onset post-transplant diabetes. The meeting time will be equivalent to those of the intervention group

The maintenance phase will last 6 months. At month 7, just as the intervention group, participants will be reminded to continue their use of the Fitbit activity tracker and that the research team will not be in contact with them for 6 months. There will be a final meeting at month 12.

Study staff will provide assistance as needed by reading questions to participants. Outcome data from both study groups will be collected at the appropriate sessions.

Retention: Text messages will be sent to participants during months when they are not attending a face-to-face session to provide encouragement and reinforcement for their participation in the study. In addition, phone calls will be made by research staff during each month to each participant to provide updates on their progress in the study as well as encouragement and support. Participants who complete the study will be allowed to keep their activity tracker.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipient at The Ohio State University Wexner Medical Center, Kidney Transplant Program
* Age 60 or older
* Received clearance from healthcare provider to participate
* Ability to speak, read, and hear English
* Possession or ready-access to a smart phone capable of accessing mobile activity tracker data
* Lacks cognitive impairment (verified by mini cognition test)
* Able to walk without an assist device (cane or walker)
* Not currently hospitalized
* Greater than 3 months post- transplant

Exclusion Criteria:

* Currently on dialysis
* Currently participating in a weight loss program
* Currently participating in a structured exercise program
* Currently wearing/using an activity tracker
* Planning to relocate out of the Columbus area in the next 6 months or less

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara O'Brien, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Kidney Transplant Program, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] O'Brien T, Russell CL, Tan A, Mion L, Rose K, Focht B, Daloul R, Hathaway D. A Pilot Randomized Controlled Trial Using SystemCHANGE Approach to Increase Physical Activity in Older Kidney Transplant Recipients. Prog Transplant. 2020 Dec;30(4):306-314. doi: 10.1177/1526924820958148. Epub 2020 Sep 10. PMID 32912051
- [Derived] O'Brien T, Russell CL, AlKahlout N, Rosenthal A, Meyer T, Tan A, Daloul R, Hathaway D. Recruitment of Older Kidney Transplant Recipients to a Longitudinal Study. Nurs Res. 2020 May/Jun;69(3):233-237. doi: 10.1097/NNR.0000000000000406. PMID 31688340

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was no pre-assignment.
Groups:
- Intervention: This arm includes participants randomize to the intervention group who will receive the combination of the SystemCHANGE & activity tracker intervention
  SystemCHANGE & Fitbit (Intervention): Study procedures include group sessions with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12. Study personnel will demonstrate proper Fitbit activity tracker use, and teach participants to sync to their smartphone and retrieve data from their Fitbit. Subjects will be called to be encouraged to increase their step goal 5% each month. Fitbit activity tracker reports will be reviewed and participants will be asked to identify what people or things influence their physical activity. Subjects will be asked what they are learning about physical activity, their contentment level with current physical activity, and if they want to make changes. Participants will continue for months, after which time there will be a final group session.
Period: Overall Study
Arm/Group | Control | Intervention
Started | 30 | 30
Completed | 23 | 23
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 7 | 7

BASELINE CHARACTERISTICS:
Population: Control group: Consented participants (n = 4) did not start the study. Intervention group: Consented participants (n= 3) did not start study. Recruitment target of 60 participants was met. Therefore, the control group had 26 participants and intervention group had 27 participants.
Groups:
- Intervention: This are includes participants randomize to the intervention group who will receive the combination of the SystemCHANGE and activity tracker intervention
  SystemCHANGE and Fitbit (Intervention): Study procedures include group sessions with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12. Study personnel will demonstrate proper Fitbit activity tracker use, and teach participants to sync to their smartphone and retrieve data from their Fitbit. Subjects will be called to encourage them to increase their step goal 5% each month. Fitbit activity tracker reports will be reviewed and participants will be asked to identify what people or things influence their physical activity. Subjects will be asked what they are learning about physical activity, their contentment level with current physical activity, and if they want to make changes..
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 11 | 15 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (4.0) | 65.7 (4.9) | 65.4 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 16 | 23
  Male | 19 | 11 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: We met our recruitment target
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 10 | 10 | 20
    White | 14 | 16 | 30
    More than one race | 2 | 0 | 2
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53
Steps per Day [Mean (Standard Deviation); unit: steps per day] — Adherence of activity tracker use was assessed by steps per day.
  steps per day | 4171 (1709) | 4432 (1865) | 4302 (1787)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 150.2 (19.05) | 141.8 (24.28) | 146 (21.66)
Diastolic Blood Pressure (mmHg [Mean (Standard Deviation); unit: mmHg] | 79.64 (10.02) | 80.16 (14.82) | 80.1 (12.4)
Heart Rate (beats per minute) [Mean (Standard Deviation); unit: beats per minute] | 74.36 (10.83) | 70.68 (10.36) | 72.62 (10.4)
Weight (pounds) [Mean (Standard Deviation); unit: pounds] | 194.4 (40.84) | 189.4 (36.3) | 191.6 (38.6)
Waist Circumference (centimeters [Mean (Standard Deviation); unit: centimeters] | 40.94 (5.13) | 40.54 (5.21) | 40.6 (5.18)
Quality of Life Physical Function [Mean (Standard Deviation); unit: scores on a scale, ranging from "0-100"] — scale ranging from 0 (lowest health) to 100 (best health)
  scores on a scale, ranging from "0-100" | 43.03 (10.07) | 41.53 (9.49) | 42.3 (9.78)
Quality of Life Mental Health [Mean (Standard Deviation); unit: scores on a scale ranging from "0 - 100"] — scale ranging from 0 (lowest health) to 100 (best health)
  scores on a scale ranging from "0 - 100" | 54.61 (9.38) | 53.68 (9.17) | 54.1 (9.2)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (5.2) | 31.1 (5.9) | 30.8 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Steps Taken Per Day by Using an Activity Tracker
Description: Steps were averaged per day.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: Descriptive statistics were used to analyze the monthly average for daily steps at 12 months.
Measure: Mean (Standard Deviation); unit: average of steps per day
Groups:
- Intervention: This are includes participants randomize to the intervention group who will receive the combination of the SystemCHANGE and activity tracker intervention
  SystemCHANGE and Fitbit (Intervention): Study procedures include group sessions with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12. Study personnel will demonstrate proper Fitbit activity tracker use, and teach participants to sync to their smartphone and retrieve data from their Fitbit. Subjects will be called to encourage them to increase their step goal 5% each month. Fitbit activity tracker reports will be reviewed and participants will be asked to identify what people or things influence their physical activity. Subjects will be asked what they are learning about physical activity, their contentment level with current physical activity, and if they want to make changes. .
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
average of steps per day
  (T2) 3months | 4710 (2628) | 5708 (3586)
  (T3) 6months | 4157 (2931) | 4981 (3028)
  (T4) 12months | 3608 (2985) | 4766 (3114)

2. Secondary Outcome: Six Minute Walk Test
Description: A section of 98 feet was marked off on a hard flat surface using two orange cones. Participants were asked to walk at a comfortable pace for 6-minutes between the cones while being timed, and the distance walked was recorded in feet.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: Mixed-effects linear regression modeling was used to model the Six Minute Walk Test as a linear combination of the fixed-effects of group (intervention vs. attention-control).
Measure: Mean (Standard Deviation); unit: Feet
Groups:
- Intervention: This are includes participants randomize to the intervention group who will receive the combination of the SystemCHANGE and activity tracker intervention.
  SystemCHANGE and Fitbit (Intervention): Study procedures include group sessions with 10-12 participants for 6 months and a 6-month maintenance phase without contact from study personnel until month 12. Study personnel will demonstrate proper Fitbit activity tracker use, and teach participants to sync to their smartphone and retrieve data from their Fitbit. Subjects will be called to encourage them to increase their step goal 5% each month. Fitbit activity tracker reports will be reviewed and participants will be asked to identify what people or things influence their physical activity. Subjects will be asked what they are learning about physical activity, their contentment level with current physical activity, and if they want to make changes.
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
Feet
  (T2) 3Months | 1142 (337.1) | 1158 (235.9)
  (T3) 6 Months | 1204 (266.6) | 1142 (295.0)
  (T4) 12 Months | 1146 (264.7) | 1120 (259.4)

3. Secondary Outcome: Resting Blood Pressure
Description: Resting blood pressure will be measured on each participant in a seated position using a Withings blood pressure cuff by the research staff. The research staff collecting the resting blood pressure reading will be a registered nurse. The research staff collecting the readings will be blinded to the study groups.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: We used mixed-effects linear regression modeling to derive estimates for the resting blood pressure.
Measure: Mean (Standard Deviation); unit: (mmHg)
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
(mmHg)
  (T2) 3 months Systolic Blood Pressure (Unit of Measure: mmHg) | 146.7 (18.61) | 140.7 (26.54)
  (T2) 3 months Diastolic Blood Pressure (Unit of Measure: mmHg) | 80.52 (12.73) | 79.52 (14.47)
  (T3) 6 months Systolic Blood Pressure (Unit of Measure: mmHg) | 142.2 (12.76) | 143.3 (19.69)
  (T3) 6 months Diastolic Blood Pressure (Unit of Measure: mmHg) | 77.20 (8.94) | 78.80 (13.10)
  (T4) 12 months Systolic Blood Pressure (Unit of Measure: mmHg) | 143.8 (16.59) | 132.2 (14.80)
  (T4) 12 months Diastolic Blood Pressure (Unit of Measure: mmHg) | 77.38 (10.21) | 74.05 (10.19)

4. Secondary Outcome: Quality of Life: Physical (Functional) and Mental (Well-being) Health"
Description: Physical and mental component scores, ranging from 0 (lowest level of health) to 100 (highest level of health), are derived from the individual items and was used as study outcomes.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: We used mixed-effects linear regression modeling to derive estimates for the quality of life.
Measure: Mean (Standard Deviation); unit: score from 0-100
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
score from 0-100
  Quality of Life (T2) 3 months Physical Function | 45.32 (7.84) | 40.37 (9.34)
  Quality of Life (T3) 6 months Physical Function | 44.69 (9.25) | 40.91 (9.97)
  Quality of Life (T4) 12 months Physical Function | 45.71 (7.93) | 40.02 (8.18)
  Quality of Life Mental Health ( T2) 3 months | 53.50 (8.03) | 54.68 (8.51)
  Quality of Life Mental Health ( T3) 6 month | 53.12 (9.87) | 51.30 (8.21)
  Quality of Life Mental Health ( T4) 12 months | 50.91 (10.69) | 51.56 (9.93)

5. Secondary Outcome: Weight (Pounds)
Description: Weight was measured without shoes and in light clothing using a digital scale.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: We used mixed-effects linear regression modeling to derive estimates for the weight.
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
pounds
  (T2) 3 months (pounds) | 193.1 (36.63) | 188.5 (37.11)
  (T6) 6 months (pounds) | 192.6 (36.06) | 186.6 (37.67)
  (T4) 12 months (pounds) | 189.0 (35.91) | 189.3 (37.17)

6. Secondary Outcome: Radial Pulse (Beats Per Minute)
Description: The research staff will obtain a radial pulse (heart rate) over a 60-second count while the participant remains seated. The research staff collecting the radial pulse reading will be a registered nurse and blinded to the study groups.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: We used mixed-effects linear regression modeling to derive estimates the resting heart rate.
Measure: Mean (Standard Deviation); unit: (beats per minute)
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
(beats per minute)
  (T3) 3 months(beats per minute) | 70.20 (12.11) | 69.08 (8.82)
  (T3) 6 months(beats per minute) | 70.20 (11.11) | 67.56 (11.30)
  (T4) 12 months(beats per minute) | 67.21 (8.20) | 66.82 (7.76)

7. Secondary Outcome: Body Mass Index (BMI)kg/m2
Description: Body mass index (BMI; kg/m2) will be calculated as [mass (lb)/ height (in)2 x 703
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: Mixed-effects linear regression modeling was used to model the BMI.
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
kg/m2
  (T2) 3 months kg/m2 | 30.3 (5.5) | 31.3 (6.1)
  (T3) 6 months kg/m2 | 29.5 (4.6) | 30.7 (6.4)
  (T4) 12months kg/m2 | 28.4 (4.4) | 29.5 (8.1)

8. Secondary Outcome: Health Outcome: Waist Circumference (cm)
Description: Waist circumference (WC) will be obtained by measuring the individual's circumference halfway between the illac crest and the lower anterior ribs with the person standing upright during expiration.
Time Frame: (T2) 3months, (T3) 6months, & (T4)12 months
Population: We used mixed-effects linear regression modeling to derive estimates for each the WC.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Intervention
Number analyzed (Participants) | 26 | 27
cm
  (T2) 3 Months (cm) | 39.76 (5.24) | 39.22 (5.00)
  (T3) 6 Months (cm) | 39.08 (4.92) | 38.68 (5.02)
  (T4) 12 Months (cm) | 38.42 (4.66) | 38.70 (5.42)

ADVERSE EVENTS:
Time Frame: No adverse events occurred over the duration which the adverse events were assessed up to 12 months.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03191630/Prot_SAP_000.pdf